CLINICAL TRIAL: NCT07112664
Title: Accuracy of Fully Guided Dental Implant Placement: A Comparative Study of Experienced vs. Novice Clinicians Using Unilateral Tooth Supported, Bilateral Tooth Supported, and Soft Tissue Supported Guides
Brief Title: Accuracy of Fully Guided Dental Implant Placement by Experienced and Novice Clinicians Using Different Surgical Guides
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abdelrahman Khalaf Eldabe (Other)
Responsible Party: Sponsor-Investigator, Abdelrahman Khalaf Eldabe, Lecturer of Oral Medicine and Periodontology , Assiut University, Assiut University
Organization: Assiut University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17-2025-00015
Record Dates: First submitted 2025-08-02; First posted 2025-08-08 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Accuracy of Fully Guided Dental Implant Placement Based on Clinician Experience and Surgical Guide Support Type
Keywords: Dental Implants, Fully Guided Surgery, Guided Implant Placement, Surgical Guide Accuracy, Implant Deviation, Dental Implantology, Digital Implant Planning

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Experienced Clinician - Bilateral Tooth-Supported Guide (Experimental): Experienced Clinician - Bilateral Tooth-Supported Guide Participants receive fully guided dental implant placement using a bilateral tooth-supported surgical guide. The procedure is performed by an experienced clinician with over 500 guided implant placements.
  Interventions: Device: Fully Guided Dental Implant Placement Using Surgical Guide
- Experienced Clinician - Unilateral Tooth-Supported Guide (Experimental): Experienced Clinician - Unilateral Tooth-Supported Guide Participants receive fully guided dental implant placement using a unilateral tooth-supported surgical guide. The procedure is conducted by an experienced clinician.
  Interventions: Device: Fully Guided Dental Implant Placement Using Surgical Guide
- Experienced Clinician - Mucosa-Supported Guide (Experimental): Participants receive fully guided dental implant placement using a mucosa-supported surgical guide. The procedure is performed by an experienced clinician with extensive experience in guided surgery.
  Interventions: Device: Fully Guided Dental Implant Placement Using Surgical Guide
- Novice Clinician - Bilateral Tooth-Supported Guide (Experimental): Participants receive fully guided dental implant placement using a bilateral tooth-supported surgical guide. The procedure is performed by a novice clinician with fewer than 20 guided implant cases and at least one year of general implant experience.
  Interventions: Device: Fully Guided Dental Implant Placement Using Surgical Guide
- Novice Clinician - Unilateral Tooth-Supported Guide (Experimental): Participants receive fully guided dental implant placement using a unilateral tooth-supported surgical guide, performed by a novice clinician.
  Interventions: Device: Fully Guided Dental Implant Placement Using Surgical Guide
- Novice Clinician - Mucosa-Supported Guide (Experimental): Participants receive fully guided dental implant placement using a mucosa-supported surgical guide. The procedure is carried out by a novice clinician under standard protocol.
  Interventions: Device: Fully Guided Dental Implant Placement Using Surgical Guide

INTERVENTIONS:
Device: Fully Guided Dental Implant Placement Using Surgical Guide — All participants will undergo fully guided dental implant placement using a 3D-printed surgical guide (tooth-supported or mucosa-supported). The surgical guide is designed and fabricated based on preoperative CBCT and intraoral scan data. Implant site preparation and fixture insertion are performed entirely through the guide using manufacturer-specific guided surgery kits.

SUMMARY:
The goal of this clinical trial is to learn how accurate fully guided dental implant placement is when performed by experienced versus novice clinicians. It will also study how different types of surgical guides affect the accuracy of implant placement.

The main questions it aims to answer are:

Does the clinician's level of experience affect how closely the dental implant matches the planned position?

Does the type of surgical guide (tooth-supported or mucosa-supported) influence implant placement accuracy?

Researchers will compare the implant accuracy across six groups based on clinician experience and guide type.

Participants will:

Undergo a fully guided dental implant procedure using a 3D-printed surgical guide

Be treated by either an experienced or a novice clinician

Receive follow-up scans to measure how accurately the implant was placed compared to the digital plan

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Clinical situation suitable for dental implant placement as judged by the examining physician or principal investigator
* Adequate soft and hard tissue conditions for implant placement
* Adequate occlusion in the implant area
* Sufficient bone volume to place the implant without bone augmentation (i.e., at least 2 mm of bone circumferentially around the implant site based on preoperative CBCT)

Exclusion Criteria:

* Major systemic diseases (e.g., uncontrolled diabetes, immunosuppressive conditions)
* Untreated or uncontrolled dental caries
* Active periodontal disease
* Requirement for bone augmentation or sinus lift in the implant area
* Current pregnancy
* Current smoker (defined as >10 cigarettes per day)
* Noncompliance or inability to follow study protocols
* Known allergies to materials used in the implant system or medications administered

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Angular Deviation | Immediately postoperative (within 1 day after implant placement)
  The angular deviation is defined as the angle (in degrees) between the long axis of the virtually planned implant and the long axis of the actual placed implant. It reflects the angular accuracy of guided implant placement.

SECONDARY OUTCOMES:
Coronal Global Deviation (CGD) | Immediately postoperative
  The linear distance (in mm) between the apical center of the planned and placed implant.
Apical Global Deviation (AGD) | Immediately postoperative
  The linear distance (in mm) between the apical center of the planned and placed implant.
Depth Deviation | Immediately postoperative
  The difference in depth (in mm) between the planned and actual implant positions along the implant's central axis.

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Asyut Governorate, Egypt